CLINICAL TRIAL: NCT03880591
Title: Baseline Assessment of Neonatal Hyperbilirubinaemia in a Cohort of New-borns in Kinshasa, Democratic Republic of Congo
Brief Title: Neonatal Hyperbilirubinaemia in the Democratic Republic of Congo
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: NEHYA
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Neonatal Screening Cards (dried blood spots)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neonatal hyperbilirubinaemia (NH) is common among healthy neonates and normally resolves within a week. Untreated pathological hyperbilirubinaemia, however, can result in long-term neurological sequelae, which compromise childhood development, or may result in perinatal death. True population-based data from middle to low-income countries are scarce and NH contribution to morbidity and mortality remains unclear. With this study the investigators aim at assessing the prevalence of neonatal hyperbilirubinaemia in a cohort of newborns in a maternity hospital in Kinshasa, the Democratic Republic of Congo, and at evaluating the possible risk factors for NH in the mother and the baby.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinaemia is common among healthy neonates and normally resolves within a week. Untreated pathological hyperbilirubinaemia, however, can result in long-term neurological sequelae, which compromise childhood development, or may result in perinatal death. Worldwide, this condition aﬀects at least 481,000 term or near term newborn babies annually, causing 114,000 deaths and more than 63,000 cases of moderate or severe disability. In high-income settings, early diagnosis and treatment in neonatal intensive care units have dramatically improved the outcome for babies at risk. However, true population-based data from middle to low-income countries are scarce and NH contribution to morbidity and mortality remains unclear. The Democratic Republic of Congo is one of the 5 countries with the highest neonatal mortality rate: 29 per 1000 live births, with an estimated 96,963 annual deaths. NH diagnosis is mostly performed by visual inspection, which is not very reliable, and it is not systematically reported in maternity records. The primary objective is to evaluate the prevalence of neonatal hyperbilirubinaemia in a cohort of in-hospital consecutive live births. The secondary objective is to evaluate the possible risk factors for NH in the mother and the baby. The results of this survey will provide essential baseline data for the community. If the frequency of the NH and severe NH in the area is higher than routinely reported, prompt and appropriate management guidelines can be put in place to improve treatment to decrease neonatal mortality and neurological disabilities.

ELIGIBILITY:
Inclusion Criteria:

* All live male or female new-borns
* Mothers of any age, willing and able to give informed consent for participation in the survey and agree to stay 72 hours in hospital after giving birth

Exclusion Criteria:

* Newborn health conditions which makes difficult to drawn a blood sample
* Newborn health conditions requiring specific care not compatible with the survey procedures

Max Age: 60 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 306 in-hospital consecutive live births
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of neonatal hyperbilirubinaemia in a cohort of newborns | 72 hours
  Number of newborns with elevation of serum bilirubin to a level requiring treatment according to consensus-based bilirubin thresholds for gestational age within 72 hours from birth (https://www.nice.org.uk/guidance/cg98/resources)

SECONDARY OUTCOMES:
Risk factors for neonatal hyperbilirubinaemia in the mother and the baby | At birth
  Prevalence of Low Birth Weight (weight at birth), Prematurity (Estimated Gestational Age), Glucose-6-Phosphate Dehydrogenase deficiency and Sickle Cell Disease (both diagnosed by DNA analysis from Neonatal Screening Card), mother - child ABO and Rh factor blood incompatibility (Beth-Vincent and agglutination test), maternal malarial infection (microscopy) and sepsis (clinically diagnosed)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Fanello, Principal Investigator — University of Oxford
Locations (1):
- Kinshasa Medical Oxford Research Unit, Kinsasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slusher TM, Zamora TG, Appiah D, Stanke JU, Strand MA, Lee BW, Richardson SB, Keating EM, Siddappa AM, Olusanya BO. Burden of severe neonatal jaundice: a systematic review and meta-analysis. BMJ Paediatr Open. 2017 Nov 25;1(1):e000105. doi: 10.1136/bmjpo-2017-000105. eCollection 2017. PMID 29637134
- [Derived] Fanello C, Lee SJ, Bancone G, Kayembe D, Ndjowo P, Badjanga B, Gornsawun G, Chotthanawathit P, Waithira N, White NJ, Onyamboko M. Prevalence and Risk Factors of Neonatal Hyperbilirubinemia in a Semi-Rural Area of the Democratic Republic of Congo: A Cohort Study. Am J Trop Med Hyg. 2023 Sep 5;109(4):965-974. doi: 10.4269/ajtmh.23-0293. Print 2023 Oct 4. PMID 37669757